CLINICAL TRIAL: NCT01625468
Title: Brief Interventions to Create Smoke-Free Home Policies in Low-Income Households
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of North Carolina, Chapel Hill (Other); The University of Texas Health Science Center, Houston (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Michelle C. Kegler, Director, Emory Prevention Research Center, & Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00056797; U01CA154282-01 (NIH)
Record Dates: First submitted 2012-05-31; First posted 2012-06-21 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Diseases
Keywords: Secondhand smoke exposure; Smoke-free homes; Smoke-free home bans
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participant receives usual care
- Intervention (Experimental): Intervention group participants receive three sets of mailed educational materials about making their home smoke-free and one coaching call.
  Interventions: Behavioral: Educational print materials and a coaching call

INTERVENTIONS:
Behavioral: Educational print materials and a coaching call — Intervention group participants receive three sets of mailed educational materials about making their home smoke-free and one coaching call.
  Arms: Intervention

SUMMARY:
The burden of tobacco use falls disproportionately on low-income populations, through high rates of primary smoking and exposure to secondhand smoke. The remarkable progress in creating smoke-free environments in the U.S. over the past two decades has left smoker's homes as one of the primary sources of exposure to secondhand smoke for both children and nonsmoking adults. Intervention research that identifies effective and practical strategies for reaching the minority of households that still allow smoking in the home has considerable potential to reduce smoke exposure, but suitable channels to reach low-income families are limited. The proposed research will develop, evaluate and disseminate a brief smoke-free homes intervention through the established national infrastructure of 2-1-1 call centers. 2-1-1 is a nationally designated 3-digit telephone exchange, similar to 9-1-1 for emergencies or 4-1-1 for directory assistance, that links callers to community-based health and social services.

The proposed research has four specific aims: 1) Conduct formative research on intervention messages and materials for promoting smoke-free homes in low-income populations, applicable to both smokers and nonsmokers as household change agents; 2) Conduct a randomized controlled trial in the Atlanta 2-1-1 service area to evaluate the efficacy of a brief intervention to create smoke-free homes among 2-1-1 callers; 3) Conduct replication studies in Houston and North Carolina 2-1-1 systems to systematically test the intervention in varied populations and tobacco control climates, and 4) Disseminate the research-tested smoke-free homes intervention through a variety of mechanisms including a national grants program to 2-1-1 systems and through the Tobacco Technical Assistance Consortium's linkages to the state and local tobacco control infrastructure in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older.
* Must speak and understand English.
* Must smoke and live with at least one other non-smoking person OR be a non-smoker who lives with a smoker(s).
* Must not have a total smoking ban in their home.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Presence of a total home smoking ban | Change from baseline in reported total home smoking bans at 3-month and 6-month follow-up

SECONDARY OUTCOMES:
Weekly secondhand smoke exposure for non-smokers | Change from baseline in reported secondhand smoke exposure for non-smokers at 3-month and 6-month follow-up
Cessation attempts (for smokers) | Change from baseline in reported cessation attempts (for smokers) at 3-month and 6-month follow-up
Number of cigarettes smokes (for smokers) | Change from baseline in reported number of cigarettes smoked (for smokers) at 3-month and 6-month follow-up
Stage of change to quit smoking (for smokers) | Change from baseline in stage of change to quit smoking (for smokers) at 3-month and 6-month follow-up
Successful cessation (for smokers) | Change from baseline in successful cessation (for smokers) at 3-month and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kegler, DrPH, Principal Investigator — Emory University
Locations (1):
- Emory University Rollins School of Public Health, Atlanta, Georgia, United States

REFERENCES:
- [Background] Kegler MC, Escoffery C, Bundy L, Berg CJ, Haardorfer R, Yembra D, Schauer G. Pilot study results from a brief intervention to create smoke-free homes. J Environ Public Health. 2012;2012:951426. doi: 10.1155/2012/951426. Epub 2012 May 17. PMID 22675374
- [Background] Berg CJ, Bundy L, Escoffery C, Haardorfer R, Kegler MC. Telephone-assisted placement of air nicotine monitors to validate self-reported smoke-free home policies. Public Health. 2013 Apr;127(4):342-4. doi: 10.1016/j.puhe.2013.01.002. Epub 2013 Mar 6. PMID 23480954
- [Background] Escoffery C, Bundy L, Carvalho M, Yembra D, Haardorfer R, Berg C, Kegler MC. Third-hand smoke as a potential intervention message for promoting smoke-free homes in low-income communities. Health Educ Res. 2013 Oct;28(5):923-30. doi: 10.1093/her/cyt056. Epub 2013 May 13. PMID 23669213
- [Result] Kegler MC, Bundy L, Haardorfer R, Escoffery C, Berg C, Yembra D, Kreuter M, Hovell M, Williams R, Mullen PD, Ribisl K, Burnham D. A minimal intervention to promote smoke-free homes among 2-1-1 callers: a randomized controlled trial. Am J Public Health. 2015 Mar;105(3):530-7. doi: 10.2105/AJPH.2014.302260. Epub 2015 Jan 20. PMID 25602863
- [Derived] Haardorfer R, Kreuter M, Berg CJ, Escoffery C, Bundy LT, Hovell M, Mullen PD, Williams R, Kegler MC. Cessation and reduction in smoking behavior: impact of creating a smoke-free home on smokers. Health Educ Res. 2018 Jun 1;33(3):256-259. doi: 10.1093/her/cyy014. PMID 29788227
- [Derived] Kegler MC, Haardӧrfer R, Berg C, Escoffery C, Bundy L, Williams R, Mullen PD. Challenges in Enforcing Home Smoking Rules in a Low-Income Population: Implications for Measurement and Intervention Design. Nicotine Tob Res. 2016 May;18(5):976-81. doi: 10.1093/ntr/ntv165. Epub 2015 Aug 5. PMID 26246049